CLINICAL TRIAL: NCT04941274
Title: A Phase I/II Study of Abemaciclib in Patients With HIV-associated and HIV-negative Kaposi Sarcoma
Brief Title: Abemaciclib in Patients With HIV-associated and HIV-negative Kaposi Sarcoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 210026; 21-C-0026
Record Dates: First submitted 2021-06-25; First posted 2021-06-28 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01-20

CONDITIONS: Kaposi Sarcoma
Keywords: Angiogenesis; AIDS; cyclin-dependent kinase; KSHV; Cell Cycle
MeSH Terms: conditions — Sarcoma, Kaposi; Acquired Immunodeficiency Syndrome | interventions — abemaciclib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1/Dose Determination/De-Escalation (Experimental): Abemaciclib (de-escalating dose)
  Interventions: Drug: Abemaciclib
- 2/Dose Expansion: Group 2a (Experimental): Abemaciclib (at optimal dose determined in dose escalation portion of the study) for up to 15 participants previously treated with at least 1 line of systemic therapy.
  Interventions: Drug: Abemaciclib
- 2/Dose Expansion: Group 2b (Experimental): Abemaciclib (at optimal dose determined in dose escalation portion of the study) for up to 10 previously untreated participants.
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Abemaciclib — An initial dose of 200 mg twice daily and at an MTD dose will be administered orally every day of each 28-day cycle.

SUMMARY:
Background:

Kaposi Sarcoma (KS) is common in people with human immunodeficiency virus (HIV) but can also occur in people who do not have HIV. KS tumors usually involve the skin, but may also involve lymph nodes, lungs, bone, and gastrointestinal tract. Researchers want to see if a drug that is currently used to treat a type of breast cancer can help.

Objective:

To find a safe dose of abemaciclib to treat KS and to see if it can shrink lesions or tumors.

Eligibility:

People ages 18 and older with KS.

Design:

Participants will be screened with some or all of the following:

Medical history

Physical exam

Blood and urine tests

Chest x-ray and/or computed tomography scans

Lung or gastrointestinal tract exam with an endoscope (a flexible instrument to examine the interior of the organ)

Medicine review

Heart function tests

KS lesion assessment

Skin sample from a KS lesion

Treatment will be given in 28-day cycles. Participants will take the study drug tablets by mouth everyday. They will keep a medicine diary. They will get the study drug until their cancer gets worse or they have unacceptable side effects.

Participants will have a study visit at the beginning of each cycle. At these visits, they will repeat some screening tests. They may have medical photographs taken of body surfaces. They may complete questionnaires about their quality of life. They may give skin and saliva samples. For skin samples, an area of skin will be numbed. A small circle of skin over an area affected by KS will be removed.

Participants will have follow-up visits for up to 2 years after treatment ends.

DETAILED DESCRIPTION:
Background:

* Kaposi Sarcoma (KS) is a multicentric angioproliferative tumor, caused by Kaposi sarcoma-associated herpesvirus, that most frequently involves the skin, but may also involve lymph nodes, lungs, bone and gastrointestinal tract. It is most common in people with HIV but may also occur in patients without a diagnosis of HIV. Patients with HIV-associated KS have worse survival than HIV-infected patients without KS.
* As it is a relapsing and remitting condition, patients with KS often require prolonged courses of cytotoxic chemotherapy and improved approaches for refractory and recurrent KS are needed to decrease morbidity among patients with KS.
* Cell cycle dysregulation is one of the hallmarks of cancer and has been developed as a therapeutic target in patients with metastatic breast cancer. Cell cycle is controlled by several proteins, including cyclin D kinases (CDKs), cyclins and retinoblastoma (Rb)-E2F signaling pathway.
* Abemaciclib is an orally available cyclin-dependent kinase (CDK) inhibitor that targets the CDK4 (cyclin D1) and CDK6 (cyclin D3) cell cycle pathways thereby inhibiting retinoblastoma (Rb) protein phosphorylation in early G1.
* KS is an endothelial tumor, and KSHV-infected endothelial cells serve as the best current model for KS as there are no good animal models for this disease. Abemaciclib was found to inhibit proliferation of KSHV-infected and uninfected human umbilical vein endothelial cells (HUVEC) at doses as low as 0.1 microM.
* Published Phase I/II studies demonstrated that abemaciclib led to clinical responses in patients with metastatic breast cancer and other tumor types, such as glioblastoma, colorectal cancer, and melanoma.
* Abemaciclib is a therapy licensed for use in metastatic breast cancer both as monotherapy and in combination with other cancer therapies and the safety and efficacy profiles of this agent are very well known. We hypothesize that abemaciclib will be well-tolerated and participants with KS who have received prior therapies will derive some clinical benefit.

Objectives:

* Phase I: To assess the safety and tolerability of abemaciclib in participants with KS
* Phase II: To assess the overall response rate (ORR) of abemaciclib of all participants and by prior KS therapy (untreated KS vs. previously treated KS), and by Stage T1 KS

Eligibility:

* Age >=18 years
* Histologically confirmed Kaposi sarcoma (KS)
* KS requiring systemic therapy, with either no prior systemic therapy or history of at least 1 prior line of systemic therapy:

  * 3 weeks from last chemotherapy
  * 3 weeks from last immunotherapy
* Measurable disease consisting of at least five measurable cutaneous KS lesions with no previous local radiation, surgical or intralesional cytotoxic therapy to these measurable lesions; or, in the absence of measurable cutaneous lesions or less than 5 lesions, evaluable KS by RECIST criteria would be required.
* ECOG Performance Status (PS) <= 2
* Participant must be willing to give informed consent.
* Participants can be HIV positive or negative.
* Antiretroviral therapy (ART) for HIV+ participants
* Participants receiving other investigational agents will not be eligible.

Design:

* This is a Phase I/II study assessing the safety and efficacy of abemaciclib in participants with previously untreated or treated KS.
* In the Phase I portion of the study, up to 18 KS participants treated with prior therapy will be enrolled in a 3+3 dose de-escalation schema using 2 dose de-escalation levels.
* Following identification of an optimal dose and schedule, an expansion phase (Phase II) will be initiated. The Phase II will involve multiple groups: up to 25 previously untreated or treated KS participants will be enrolled; and, up to 23 KS participants with Stage T1 disease.
* Abemaciclib will be administered as an oral planned starting dose of 200 mg twice daily (in the morning and evening) without regard to meals. Abemaciclib will be given continuously; one cycle equals 28 days.
* Participants will receive therapy until optimal tumor response, unacceptable toxicity, the participant s request to discontinue therapy, or Principal Investigator (PI) decision. Participants with disease progression will have the option of an additional 12 weeks of treatment, if the PI feels that they are deriving clinical benefit.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have Kaposi sarcoma confirmed by the Laboratory of Pathology, NCI
* Measurable disease as follows:

  * All participants in Groups 1, 2a, or 2b should have at least five measurable cutaneous KS lesions per AIDS Clinical Trials Group Oncology Committee (ACTG) criteria with no previous local radiation, surgical or intralesional cytotoxic therapy that would prevent response assessment for that lesion.
  * Measurable disease by the criteria proposed by the AIDS Clinical Trials Group Oncology Committee.
  * Participants in Group 3 must have Stage T1 KS with at least five measurable cutaneous KS lesions per ACTG criteria and/or evaluable disease per RECIST criteria.
* Participants may be HIV positive or negative.
* Participants must be able to swallow oral medications
* For all groups, participants must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count >1,000/mcL
  * Platelets >75,000/mcL
  * Hemoglobin >= 8gm/dL
  * Total bilirubin <= 1.5 upper limit of normal unless the participant is receiving a protease inhibitor known to be associated with increased bilirubin (e.g. atazanavir), in which case total bilirubin <= 7.5 mg/dL with direct fraction <= 0.7
  * AST/ALT <3 X institutional upper limit of normal
  * Creatinine within normal institutional limits OR
  * Creatinine clearance >45 mL/min/1.73 m^2 as estimated by either Cockroft-Gault or 24-hour urine collection for participants with creatinine levels above institutional normal
  * Cardiac ejection fraction > 45% by echocardiogram
* Prior Treatment as follows:

  * For Phase I: Participants must have received at least 1 prior line of systemic therapy for KS with either plateau in response, progressive disease, or inadequate response to treatment. Previous local therapy or radiation is not considered systemic therapy.
  * For Phase II: Group 2a: Individuals must have received at least 1 prior line of systemic therapy for KS with either plateau in response, relapsed disease, progressive disease, or inadequate response to treatment
  * For Phase II: Group 2b: Individuals have not received prior systemic therapy for KS. Previous local therapy or radiation is not considered systemic therapy.
* For Phase II: Group 3: Evidence of Stage T1 KS with either a) edema or ulcerated KS and/or b) extensive oral KS and/or c) visceral KS involvement
* Age >18 years
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) <= 2 (Karnofsky >= 60%.
* Human immunodeficiency virus (HIV)-infected individuals on effective anti-retroviral therapy are eligible for this trial.
* Willingness to adhere to ART
* All participants must have received ART for 8 weeks prior to enrollment, with no evidence of KS improvement over the most recent 4 weeks
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. Participants with HCV infection who are currently on treatment are eligible if they have an undetectable HCV viral load.
* No uncontrolled severe concurrent bacterial, viral, or fungal infections.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* Contraception requirements as follows:

  * Participants of child-bearing potential (IOCBP) must agree to use a highly effective method of contraception (e.g., intrauterine device [IUD], hormonal, surgical sterilization, abstinence) prior to study entry, for the duration of study participation, and for up to 4 months after completion of abemaciclib administration
  * Participants able to father a child must with partners of childbearing potential agree to use an effective method of contraception (barrier, surgical sterilization, abstinence) for the duration of the study treatment for up to 4 months after completion of abemaciclib

administration. Individuals with partners of childbearing potential should ask their partners to be on an effective birth control (hormonal, IUD, surgical sterilization).

* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the nursing person with abemaciclib, nursing should be discontinued if the nursing person is treated with abemaciclib.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have had chemotherapy or immunotherapy within 3 weeks prior to entering the study.
* Participants who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and enrollment.
* Participants who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia or neuropathy.
* Participants who are receiving any other investigational agents.
* History of severe allergic reactions attributed to compounds of similar chemical or biologic composition to CDK inhibitor.
* Participants receiving any medications or substances that are strong/moderate inhibitors of CYP3A4 are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product.
* Serious and/or uncontrolled severe intercurrent illness that in the judgement of the investigator would preclude participation in the study.
* No active KSHV-associated multicentric Castleman disease, KSHV-associated inflammatory cytokine syndrome or primary effusion lymphoma.
* Psychiatric illness/social situations that would limit adherence with study requirements.
* Pregnancy
* Prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the regimen are eligible for this trial
* Participants with interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
safety and tolerability of abemaciclib | 28 days
  The fraction of patients with toxicity noted at each dose level will be reported by grade and type of toxicity identified.
overall response rate | every 3 cycles until completion of therapy, then every 3 months for 6 months, then every 6 months for 2 years, then annually for 2 years
  Percentage of patients with the best overall response of CR or PR to therapy

SECONDARY OUTCOMES:
KS response to abemaciclib | every 3 cycles from cycle 2 until completion of therapy, then every 3 months for 6 months, then every 6 months for 2 years, then annually for 2 years
  Staging and response to abemaciclib for KS by the evaluation of number, size, nodularity, and color of lesions.
duration of response | every 3 cycles until completion of therapy, then every 3 months for 6 months, then every 6 months for 2 years, then annually for 2 years
  The time criteria are met for CR or PR (whichever is recorded first) until the first date that patient no longer qualifies as a PR
Progression free survival | every 3 cycles until completion of therapy, then every 3 months for 6 months, then every 6 months for 2 years, then annually for 2 years
  Duration of time from the start of the treatment until time of disease relapse from PR, disease progression, or death, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Ramya M Ramaswami, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@Requests for all collected IPD data from clinical trials, conducted under a binding collaborative agreement between NCI/DCTD and a pharmaceutical/biotechnology company, that are not under DSMB monitoring must be in compliance with the terms of the binding collaborative agreement and must be approved by NCI/DCTD and the Pharmaceutical Collaborator (i.e., the NCI ETCTN Director in conjunction with the NCI/DCTD Regulatory Affairs Branch)

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2021-C-0026.html